CLINICAL TRIAL: NCT02918526
Title: Hemodynamic Study With Pressure Recording Analytical Method (PRAM) of the Cardiovascular Response to the Positioning of the Extraglottic Device in Gynecological Surgery
Brief Title: Hemodynamic Study With PRAM of the Cardiovascular Response to the Positioning of the Extraglottic Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Alessandro Di Filippo, Medical Doctor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOUCareggi
Record Dates: First submitted 2016-09-24; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Intubation Complication; Hemodynamic Instability
Keywords: Laryngeal masks
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laryngeal Mask (Experimental): laryngeal mask (LMA)
  Interventions: Device: airway management
- Oro Tracheal Intubation (Active Comparator): oro tracheal intubation
  Interventions: Device: airway management

INTERVENTIONS:
Device: airway management — airway management with Laryngeal Mask or Oro Tracheal Intubation

SUMMARY:
The purpose of the study will be to record the hemodynamic response measured by traditional methods (non-invasive blood pressure and ECG) and Pressure Recording Analytical Method in patients undergoing laryngeal mask placement compared with the hemodynamic response measured in patients undergoing laryngoscopy and tracheal intubation for performing surgery in gynecological area and assess the differences with the two methods.

DETAILED DESCRIPTION:
Introduction Laryngoscopy and tracheal intubation may cause significant hemodynamic changes in the patient and induce cardiovascular complications.

Numerous studies have sought methods to reduce this risk (1-5). The extraglottic not involving either laryngoscopy or their passage through the vocal cords, have proven protective of the possible cardiovascular complications resulting from the placement of respiratory prosthesis (6,7).

Measurements of hemodynamic changes resulting from the procedures for airway management with extraglottic have not previously been carried out.

The MostCare (Vytech, Vygon Italia srl, Padova, Italy) is a monitor provided for more than 10 years at the obstetric gynecological anesthesia unit able to evaluate the hemodynamic changes in a patient based on the Pressure Recording Analytical Method (PRAM).

This is a measurement method of the cardio-circulatory performance of a patient that does not require calibration and / or insertion of a pre-estimated data because the method of analysis of the wave form of the arterial pressure is developed completely a priori (8). The measurement derives from the simultaneous analysis of the components of a pulsatile flow and the continuous flow as a ratio between the area under the curve of the pulsatile portion of the systolic pressure and the characteristic impedance Z (t). The PRAM method has proven effective in many clinical settings (9).

The Medical Device (DM) will be used in accordance with the indications of use for which it has acquired the CE mark. A morphology detection system linked to high blood pressure curve detected through non-invasive Masimo oximetry system supplied to the Hospital will be used Purpose of the study The purpose of the research will be to record the hemodynamic response measured by traditional methods (non-invasive blood pressure and ECG) and PRAM method in patients undergoing placement laryngeal mask compared with the hemodynamic response measured in patients undergoing laryngoscopy and tracheal intubation for performing surgery in gynecological area and assess the differences with the two methods

Methods This will be a prospective observational study. Data will be collected from all consecutive patients undergoing general anesthesia for gynecologic surgery for a period of 3 months or until the minimum number of 94 patients (see section statistical analysis).

In the operating room the patient will undergo to active pre-warming with hot air, peripheral venous cannulation and premedication with midazolam 0,04 mg/kg, and fentanyl 1.5 mcg/kg body weight. After the positioning of the standard monitoring systems (ECG, Non-Invasive Blood Pressure, Pulseoximetry, Neuromuscular Transmission), the signal from the Pulseoximetry will also be analyzed by the MostCare monitoring system that allows to apply the measuring method PRAM noninvasively.

After 3 minutes of high flows O2, propofol 2 mg/kg body weight and rocuronium 0.9 mg/kg body weight will be administered sequentially to the patient. Anesthesia will be maintained with propofol continuous infusion (9-12 mg/kg body weight /hour) and remifentanil continuous infusion (0.2 mcg/kg body weight /minute ). At the disappearance of the adductor muscle response to electrical stimulation of the thumb "Train of four" (TOF) applied to the ulnar nerve the positioning maneuver of the respiratory device will be performed:

* with direct laryngoscopy in the case of endotracheal intubation
* with direct insertion in the case of laryngeal mask placement. Proper placement will be evaluated by chest auscultation, spirometry and analysis of the concentration and the carbon dioxide curve in exhaled gases.

The data obtained from the PRAM and the usual monitoring will be recorded on a special sheet by an outside observer.

In the case of failed positioning of the respiratory device, the procedure will be repeated and in case of further failure will proceed as indicated by national and hospital guidelines (10), but the patient will still be excluded from the study ..

The choice of the respiratory device will depend on the type of intervention scheduled in the operating program.

The hemodynamic and monitoring data will be recorded every minute for 5 minutes for each patient.

The study duration will be 3 months (or in any case until reaching the minimum number of 94 cases).

The patients will be divided, retrospectively, in two groups according to the type of device used for airway management.

The two groups will be compared on the basis of age and anthropometric parameters. An analysis of the hemodynamic response of the two groups of patients to the positioning of the respiratory device will then conduct.

Statistical analysis A recent study (11), that analyzed the cardiac index changes in response to tracheal intubation with laryngoscope Mcintosh in comparison to the video laryngoscope laryngoscopy, showed a difference of 1 L/min/m2 (from 3.1±0.6 to 4.3±1.4 with laryngoscope McIntosh vs 3.0±0.3 to 3.2 ± 1.1 with videolaryngoscope).

Therefore, to test the hypothesis that the cardiac index difference using the airway management with traditional intubation compared to the use of the laryngeal mask is greater than or equal to 1 L/min/m2, having fixed the first type error to the 5% and the study power to 80%, it is possible to calculate that the sample size needed for a one-tailed test is represented by 47 patients per group.

The average of the data collected in each group of patients will be compared with Student's t test.

Expected results To verify, in two of homogeneous population groups for anthropometric and clinical data, the least impact on the cardiovascular system produced by the placement of laryngeal mask compared to that induced by endotracheal intubation with conventional laryngoscopy taking advantage of non-invasive hemodynamic monitoring system of the pulse oximetry MostCare (methodology PRAM) ever tested in this field.

Also to check the hemodynamic impact of any repeated attempts to both of the above maneuvers for airway management.

Ownership of the results will be accredited by the principal investigator on behalf of the AOU Careggi and the University of Florence as headings of him which has neither received nor will receive any fee for the conduct of the study.

ELIGIBILITY:
Inclusion criteria:

* Patients scheduled for elective gynecological surgery under general anesthesia
* Age >18 <50 years
* Presence of informed consent in the clinical record
* Belonging to risk classes ASA 1 - ASA 2

Exclusion criteria:

* Hypertension
* Heart failure
* Treatment with beta blockers, Ca channel blockers, antihypertensives, vagolytic
* Hypo/hyperthyroidism and its treatment
* Adrenal insufficiency and its treatment
* Autonomic neuropathy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac Index (L/min/m2) | for 5 minutes after induction of anesthesia
  Cardiac Index (L/min/m2) measured with Pulse Recording Analytic Method

SECONDARY OUTCOMES:
Heart rate (bpm) | for 5 minutes after induction of anesthesia
Blood pressure (mmHg) | for 5 minutes after induction of anesthesia
Cardiac Output (CO) (L/min) | for 5 minutes after induction of anesthesia
Stroke Volume (SV) (ml/beat) | for 5 minutes after induction of anesthesia
Stroke Volume Index (SVI) (ml/beat /m2) | for 5 minutes after induction of anesthesia
Systemic Vascular Resistance (SVR) (dynes•s /cm5) | for 5 minutes after induction of anesthesia
Cardiac Cycle Efficiency (CCE) (a dimensional value) | for 5 minutes after induction of anesthesia
Cardiac Power Output (CPO) (W). | for 5 minutes after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Filippo, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Efe EM, Bilgin BA, Alanoglu Z, Akbaba M, Denker C. Comparison of bolus and continuous infusion of esmolol on hemodynamic response to laryngoscopy, endotracheal intubation and sternotomy in coronary artery bypass graft. Braz J Anesthesiol. 2014 Jul-Aug;64(4):247-52. doi: 10.1016/j.bjane.2013.07.003. Epub 2013 Oct 25. PMID 24998108
- [Background] Lee SY, Min JJ, Kim HJ, Hong DM, Kim HJ, Park HP. Hemodynamic effects of topical lidocaine on the laryngoscope blade and trachea during endotracheal intubation: a prospective, double-blind, randomized study. J Anesth. 2014 Oct;28(5):668-75. doi: 10.1007/s00540-014-1812-z. Epub 2014 Mar 12. PMID 24619576
- [Background] Daabiss M, Hashish M. Effects of lornoxicam on the hemodynamic and catecholamine response to laryngoscopy and tracheal intubation. Eur J Clin Pharmacol. 2011 Aug;67(8):783-6. doi: 10.1007/s00228-011-1017-4. Epub 2011 Mar 3. PMID 21369950
- [Background] Min JH, Chai HS, Kim YH, Chae YK, Choi SS, Lee A, Choi YS. Attenuation of hemodynamic responses to laryngoscopy and tracheal intubation during rapid sequence induction: remifentanil vs. lidocaine with esmolol. Minerva Anestesiol. 2010 Mar;76(3):188-92. PMID 20203546
- [Background] Sun HL, Wu TJ, Ng CC, Chien CC, Huang CC, Chie WC. Efficacy of oropharyngeal lidocaine instillation on hemodynamic responses to orotracheal intubation. J Clin Anesth. 2009 Mar;21(2):103-7. doi: 10.1016/j.jclinane.2008.06.028. PMID 19329013
- [Background] Perello-Cerda L, Fabregas N, Lopez AM, Rios J, Tercero J, Carrero E, Hurtado P, Hervias A, Gracia I, Caral L, de Riva N, Valero R. ProSeal Laryngeal Mask Airway Attenuates Systemic and Cerebral Hemodynamic Response During Awakening of Neurosurgical Patients: A Randomized Clinical Trial. J Neurosurg Anesthesiol. 2015 Jul;27(3):194-202. doi: 10.1097/ANA.0000000000000108. PMID 25121397
- [Background] Agrawal G, Agarwal M, Taneja S. A randomized comparative study of intraocular pressure and hemodynamic changes on insertion of proseal laryngeal mask airway and conventional tracheal intubation in pediatric patients. J Anaesthesiol Clin Pharmacol. 2012 Jul;28(3):326-9. doi: 10.4103/0970-9185.98325. PMID 22869938
- [Background] Romano SM, Pistolesi M. Assessment of cardiac output from systemic arterial pressure in humans. Crit Care Med. 2002 Aug;30(8):1834-41. doi: 10.1097/00003246-200208000-00027. PMID 12163802
- [Background] Scolletta S, Romano SM, Biagioli B, Capannini G, Giomarelli P. Pressure recording analytical method (PRAM) for measurement of cardiac output during various haemodynamic states. Br J Anaesth. 2005 Aug;95(2):159-65. doi: 10.1093/bja/aei154. Epub 2005 May 13. PMID 15894561
- [Background] Petrini F, Accorsi A, Adrario E, Agro F, Amicucci G, Antonelli M, Azzeri F, Baroncini S, Bettelli G, Cafaggi C, Cattano D, Chinelli E, Corbanese U, Corso R, Della Puppa A, Di Filippo A, Facco E, Favaro R, Favero R, Frova G, Giunta F, Giurati G, Giusti F, Guarino A, Iannuzzi E, Ivani G, Mazzon D, Menarini M, Merli G, Mondello E, Muttini S, Nardi G, Pigna A, Pittoni G, Ripamonti D, Rosa G, Rosi R, Salvo I, Sarti A, Serafini G, Servadio G, Sgandurra A, Sorbello M, Tana F, Tufano R, Vesconi S, Villani A, Zauli M; Gruppo di Studio SIAARTI "Vie Aeree Difficili"; IRC e SARNePI; Task Force. Recommendations for airway control and difficult airway management. Minerva Anestesiol. 2005 Nov;71(11):617-57. No abstract available. English, Italian. PMID 16278626
- [Background] Abdelgawad AF, Shi QF, Halawa MA, Wu ZL, Wu ZY, Chen XD, Yao SL. Comparison of cardiac output and hemodynamic responses of intubation among different videolaryngoscopies in normotensive and hypertensive patients. J Huazhong Univ Sci Technolog Med Sci. 2015 Jun;35(3):432-438. doi: 10.1007/s11596-015-1449-7. Epub 2015 Jun 14. PMID 26072085